CLINICAL TRIAL: NCT01836705
Title: Effect of 14-day Repeated Oral Doses of SAR302503 on Ventricular Repolarization, Compared to 1-day Placebo in Adult Patients With Refractory Solid Tumors
Brief Title: Effect of SAR302503 on ECG Activity in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TES13519; 2012-005642-38 (EudraCT Number); U1111-1115-7323 (Other: UTN)
Record Dates: First submitted 2013-04-17; First posted 2013-04-22 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2014-06

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — fedratinib; Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-sequence (Experimental): SAR302503 Placebo (1 day)-SAR302503 (500 mg, oral, qd, 14 days)
  Interventions: Drug: SAR302503 (TG101348); Drug: Placebo SAR302503; Drug: Panolosetron

INTERVENTIONS:
Drug: SAR302503 (TG101348) — Pharmaceutical form:capsule
  Route of administration: oral
Drug: Placebo SAR302503 — Pharmaceutical form:capsule
  Route of administration: oral
Drug: Panolosetron — Pharmaceutical form:solution
  Route of administration: intravenous
  Other Names: Aloxi®

SUMMARY:
Primary Objective:

- To assess the effect of SAR302503 (500 mg) administered as 14-day repeated doses on the QTcF interval compared to 1-day placebo in patients with advanced solid tumors.

Secondary Objectives:

* To assess the effect of SAR302503 administered as 14-day repeated doses on heart rate (HR), QT, QTcB, and QTcN, PR and QRS compared to placebo.
* To assess the clinical and laboratory safety of SAR302503
* To document the plasma concentrations of SAR302503 at the time of ECG investigation.
* To explore the Pharmacokinetic/Pharmacodynamic relationship between SAR302503 concentration and QTcF
* To explore antitumor activity

DETAILED DESCRIPTION:
Total 7-10 weeks if not progressing to Segment 2. Segment 2 will be additional in 28-day cycles.

ELIGIBILITY:
Inclusion criteria :

- Histologically or cytologically confirmed advanced solid malignancy that is metastatic or unresectable, and for which standard curative measures do not exist

Exclusion criteria:

* Prior history of torsades de pointe, or congenital long QT syndrome.
* Conditions with screening ECG in which repolarization is difficult to interpret, or showing significant abnormalities. This includes, but is not limited to: High degree atrioventricular (AV) block, pacemaker, atrial fibrillation or flutter
* Screening ECG with QTc B or QTc F ≥480 msec (within 8 days of Day-1)
* Significant hypokalemia at screening (K+ <3.5 mmol/L) (within 8 days of Day-1)
* Significant hypomagnesemia at screening and inclusion (Mg++ <0.7 mmol/L) (within 8 days of Day -1)
* Patient receives (and cannot discontinue), or is scheduled to receive, a concomitant treatment known to carry a risk of both QT prolongation and torsade de pointe for 2 weeks before Day 1 and for the duration of Segment 1
* Absence of completion of all prior chemotherapy, biological therapy, hormonal therapy, targeted non-cytotoxic therapy ≥3 weeks; and radiotherapy ≥2 weeks prior to inclusion.
* Patients with uncontrolled brain metastases or primary brain tumor. Patients with brain metastasis are considered eligible if the patient has not received radiation therapy for brain metastasis within 2 weeks of enrollment and has been on a stable dose of steroids for ≥ 2 weeks.
* Participation in any study of an investigational agent (drug, biologic, device) within 30 days prior to initiation of study drug, unless during non-treatment phase.
* Anticipation of need for a major surgical procedure or radiation therapy during the study treatment.
* Concurrent treatment in another clinical trial or with any other cancer therapy including chemotherapy, biological therapy, hormonal therapy, radiotherapy, chemoembolization, cryotherapy, targeted non-cytotoxic therapy or patients planning to receive these treatments during the study.
* Inadequate organ function as defined by:
* Absolute neutrophil count (ANC) <1.5 X 10^9/L
* Platelet count <100 X 10^9/L
* Hemoglobin: <9 g/dL
* Serum creatinine >1.5 x the upper limit of normal (ULN)
* Serum amylase or lipase >1.5 x ULN
* Total bilirubin >1.5 x ULN
* Aspartate aminotransferase or alanine aminotransferase ≥2.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) >2 at study entry.
* Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
* Ongoing or recent history (within 3 months of Day 1 Segment 1) of clinically significant dysrrhythmia.
* Patients taking a beta blocker within 7 days to Day 1 Segment 1 and during Segment 1
* Other concurrent serious illness or medical condition, including active infection or HIV disease.
* Patients with known active (acute or chronic) Hepatitis A, B, C, and hepatitis B and or C carriers. Prior history of chronic liver disease.
* Patients with history of partial or total gastrectomy, or, if in the opinion of the investigator, have any other disorder that would inhibit absorption of oral medications.
* Any severe acute or chronic medical, neurological, or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with interpretation of study results and, in the Investigator's opinion, would make the patient inappropriate for entry into this study.
* Contra-indications for palonosetron.
* Use of drugs or herbal agents known to be at least moderate inhibitors or inducers of CYP3A4, sensitive CYP3A4 substrate, or CYP3A4 substrate with narrow therapeutic index, within 2 weeks of Day 1 and during study.
* Concomitant treatment with H2-blockers is not allowed within 7 days prior to Day 1 Segment 1 and during entire study.
* Known hypersensitivity to any excipients in IMP formulations.
* Pregnant or lactating females
* Women of childbearing potential, unless using effective contraception (other than oral contraceptives) while on study drug. Men who partner with a woman of childbearing potential, unless they agree to use effective contraception while on study drug

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
QTc Friderica (QTcF) parameter | 16 days

SECONDARY OUTCOMES:
Electrocardiographic parameters (Heart Rate) | 16 days
Electrocardiographic parameters (QT) | 16 days
Electrocardiographic parameters (QTcBazett) | 16 days
Electrocardiographic parameters (QTcN) | 16 days
Electrocardiographic parameters (PR interval) | 16 days
Electrocardiographic parameters (QRS interval) | 16 days
Anti-tumor activity | 16 or more days
Number of participants with Adverse Events | 16 or more days
Pharmacokinetic parameter: Cmax, AUC0-24, Tmax, Tmax, Ctrough | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- United States (8):
  - Investigational Site Number 840003, Los Angeles, California
  - Investigational Site Number 840007, Augusta, Georgia
  - Investigational Site Number 840002, Detroit, Michigan
  - Investigational Site Number 840001, St Louis, Missouri
  - Investigational Site Number 840004, Cincinnati, Ohio
  - Investigational Site Number 840005, Philadelphia, Pennsylvania
  - Investigational Site Number 840006, San Antonio, Texas
  - Investigational Site Number 840008, San Antonio, Texas
- Belgium (2):
  - Investigational Site Number 056001, Brussels
  - Investigational Site Number 056002, Ghent

REFERENCES:
- [Derived] Ogasawara K, Xu C, Yin J, Darpo B, Carayannopoulos L, Xue H, Palmisano M, Krishna G. Evaluation of the Potential for QTc Prolongation With Repeated Oral Doses of Fedratinib in Patients With Advanced Solid Tumors. Clin Pharmacol Drug Dev. 2021 Apr;10(4):366-375. doi: 10.1002/cpdd.850. Epub 2020 Jul 16. PMID 32673446